CLINICAL TRIAL: NCT00006420
Title: Study of Trends of Cardiovascular Disease in a Metropolitan Area.
Brief Title: Minnesota Heart Survey - Mortality and Morbidity
Acronym: MHS
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 936; R01HL065755 (NIH)
Record Dates: First submitted 2000-10-26; First posted 2000-10-27 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Death, Sudden, Cardiac
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Death, Sudden, Cardiac

GROUPS / COHORTS (1):
- Observational, no interventions

SUMMARY:
To continue surveillance of coronary heart disease (CHD) mortality and morbidity in the seven county metropolitan Minneapolis/St. Paul (Twin Cities) areas.

DETAILED DESCRIPTION:
BACKGROUND:

The Minnesota Heart Survey (MHS) is among the few population-based longitudinal studies to monitor and explain trends in coronary heart disease (CHD) mortality and morbidity, the leading cause of death and disability in the United States. It encompasses a large and well-defined community, the Minneapolis/St. Paul (Twin Cities) metropolitan area of Minnesota, comprising a population of 2.3 million (1990 census) For almost two decade the Minnesota Heart Survey has made contributions to understanding 1) the components of the decline of coronary heart disease mortality including incidence rate, hospitalized attach rate, case fatality, and population levels of CHD risk factors; and 2) the methodology of disease surveillance in a time when classification and diagnostic technologies are constantly changing.

DESIGN NARRATIVE:

The Minnesota Heart Survey continues surveillance of coronary heart disease (CHD) mortality and morbidity in the seven county metropolitan Minneapolis/St. Paul (Twin Cities) areas through the year 2002. The study will also monitor trends in acute myocardial infarction (AMI), evaluate the effect on AMI diagnosis of the widespread use of new biomarkers (troponins), perform a validation study to the previous standard, and evaluate out-of-hospital sudden cardiac death (SCD) through an autopsy study

A combination of different techniques will be used for surveillance. CHD deaths will be obtained from death certificate data from the Minneapolis Department of Public Health. Census data will be used to construct the appropriate denominators. A major focus is based on in-hospital CHD morbidity and mortality. Data from the Minnesota Hospital and Health Care Partnership, which originally receives data from 22 of the 23 area hospitals, will be used to identify and validate acute myocardial infarction (AMI) cases. Census data will again be used to obtain the appropriate denominators. An important issue in assessing time trends in hospitalized AMI attack rate is the changing definitions used to identify cases over time. A specific issue in this regard is the increasing use of troponin levels that are more sensitive than previously used CKMB levels to identify cases. Thus, a validation study will be conducted comparing these two methodologies on the same subjects. The goal of the study is to obtain correction factors so that time trends in AMI attack rates are not influenced by differences in diagnostic criteria.

A new important area of investigation is that of out of-hospital sudden cardiac deaths (SCD). Autopsy studies of 100 cases per year (about 300 total) will be conducted to describe risk factors for SCD. In addition, comparisons will be made between a control group of 600 persons in the risk factor study.

.

ELIGIBILITY:
No eligibility criteria

Ages: 30 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Cardiovascular, morbidity and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Russell Luepker — University of Minnesota

REFERENCES:
- [Background] Lin JC, Apple FS, Murakami MM, Luepker RV. Rates of positive cardiac troponin I and creatine kinase MB mass among patients hospitalized for suspected acute coronary syndromes. Clin Chem. 2004 Feb;50(2):333-8. doi: 10.1373/clinchem.2003.026708. Epub 2003 Dec 11. PMID 14670826